CLINICAL TRIAL: NCT06306664
Title: Effect of Two Different Modes of Polarized Polychromatic Non-coherent Light Therapy on Jumper's Knee
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Shahien, physiotherapist specialist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT.REC/012/004881
Record Dates: First submitted 2024-02-25; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Jumper's Knee
Keywords: Polarized Polychromatic Non Coherent Light (Bioptron)

STUDY DESIGN:
Who Masked: Participant
Masking Description: double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): the patients will receive green filter of bioptron light therapy and conventional treatment((ice application+ exercise program)) for jumper knee three times a week for four weeks.
  Interventions: Device: Bioptron
- Group B (Experimental): the patients will receive yellow filter of bioptron light therapy and conventional treatment for jumper knee three times a week for four weeks.
  Interventions: Device: Bioptron
- Control group (Placebo Comparator): the patients will receive conventional treatment (ice application+ exercise program) for jumper knee three times a week for four weeks.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Device: Bioptron — Bioptron safely treats arthritis, neck & back pain by stimulating blood circulation, reducing inflammation and relieving muscle spasms. For just ten minutes per day, our life-transforming technology offers the highest levels of pain relief by reaching deep into joints, muscles and ligaments.
  Other Names: Polarized Polychromatic Non-Coherent Light; Hyperlight
  Arms: Group A; Group B
Other: Placebo Comparator — Patients will receive ice application+Exercises program designed for jumper knee
  Arms: Control group

SUMMARY:
The purposes of this study are:

1. To examine the combined effects of Yellow CPPNLT and conventional treatment on pain intensity, pain pressure threshold, functional disability, and muscle strength in athletic jumper knee.
2. To examine the combined effects of Green CPPNLT and conventional treatment on pain intensity, pain pressure threshold, functional disability, and muscle strength in athletic jumper knee.

3 3- To compare between the effects of Yellow CPPNLT and Green CPPNLT on pain intensity, pain pressure threshold, functional disability, and muscle strength in athletic jumper knee.

DETAILED DESCRIPTION:
Jumper's knee is an overuse injury of the tendon that alters the knee due to repeated stress of activities. Symptoms include pain in the front of the knee. The tears are typically caused by accumulated stress on the patellar or quadriceps tendon. As the name implies, the condition is common in athletes from jumping sports, where there is a high demand for the speed and power of leg extensors. These sports often lead to high eccentric quadriceps loadings, such as volleyball, track (long and high jump), basketball, long-distance running, and skiing. The prevalence of jumper knee is not well examined so far. For non-elite adult athletes the prevalence varies between 14.4% and 2.5% for different sports.Only 2.4% of adolescent professional soccer players sustain PT. However, knee pain, focal tenderness or even acute episodes of PT have a major impact on each player's development, time off the pitch, and career.Bioptron was used for treatment of arthritis, neck&back pain by stimulating blood circulation, reducing inflammation and relieving muscle spasm. There are some studies that have discussed the extent of the effect of the Bioptron Light Therapy on musculoskeletal disorders such as; rotator cuff tendinitis, tennis elbow, carpal tunnel syndrome, acute patellar tendinopathy and acute ankle sprain. There is a lack of the evidence of the clinical guidelines of patellar tendinitis. Up to our knowledge, there is no clear recommendation about efficiency of different colors of Bioptron light therapy on jumper knee. So; this study will be conducted to determine efficiency of yellow and green colors of polychromatic non-coherent light. Sixty subjects will participate in this study and will be divided randomly into three equal groups.Group A (Study group): Will receive green filter of bioptron light therapy and conventional treatment for jumper knee,group B (Study group): Will receive yellow filter of bioptron light therapy and conventional treatment for jumper knee and group C (Control group): Will receive conventional treatment (ice application+ exercise program) for jumper knee.

ELIGIBILITY:
Inclusion Criteria:

* History of Patellar tendinitis and anterior knee pain.
* Age will be ranged from 15 to 35 years.
* Both genders.
* The onset of pain for over 3 months.

Exclusion Criteria:

* Knee surgery within the previous 6 months.
* Chronic joint diseases.
* Corticosteroid injection in the patellar tendon within the previous 3 months.
* Use of drugs 48 hours previously (e.g., NSAIDs).
* Any other concomitant treatment for PT.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11-29 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain (Visual analogue scale). | Visual analogue scale will be investigated at baseline and after the treatment period of 4 weeks.
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. The VAS score for grading of pain consists of a 10 centimeters (cm) line with 10 mm (0.01 cm) to each point of the scale and two end-points representing no pain and worst possible pain.
pain intensity (Pressure algometry) | Pressure algometry will be investigated at baseline and after the treatment period of 4 weeks.
  Pressure pain threshold will be measured with algometry test FPX25 using 1-cm2 rubber tip on the knee extensors.10, 11 pressures will be applied slowly until the participant first feels the pain and response by saying stop there.
Disability questionnaire (Victorian institute of sport assessment-patella). | The VISA-P questionnaire will be investigated at baseline and after the treatment period of 4 weeks.
  The VISA-P, formerly known as the Victorian institute of sport assessment -patella Questionnaire, The VISA-P is questionnaire that assesses symptoms, simple tests of function, and the ability to play sports.
Muscle strength (Hand held dynamometer) | The Lafayette hand held dynamometer will be investigated at baseline and after the treatment period of 4 weeks.
  The subjects will be positioned in sitting on chair and we will apply resistance when performing the dynamometer on patients and they will try to make maximal effort against resistance and we will record the change of length or resistance.

OTHER OUTCOMES:
Muscle strength and endurance ( Biodex-Isokinetic Dynamometer) | The Isokinetic dynamometer will be investigated at baseline and after the treatment period of 4 weeks.
  The subjects will be positioned in sitting on isokinetic chair and we will ask the subjects to perform maximal knee extension and we will record the change of muscle power or endurance

CONTACTS AND LOCATIONS:
Overall Officials: Adel R Ahmed, PHD, Study Director — Cairo University
Locations (1):
- Physical Therapy, Giza, Dokki, Egypt